CLINICAL TRIAL: NCT06406907
Title: Effects of Short Duration Blood Flow Restriction Training on Musculoskeletal and Performance Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: REC/PhD/011104 Saad Rauf
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Blood Flow Restriction Training
Keywords: Blood flow restriction; Surface EMG; Reactive strength index; Abdominal muscles
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- High Frequency Blood Flow Restriction Training Group (Experimental): Subjects allocated to this group performed squat exercise 6 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM.
  Interventions: Other: High Frequency Blood Flow Restriction Training Group
- Low Frequency Blood Flow Restriction Training Group (Experimental): Subjects allocated to this group performed squat exercise 3 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM.
  Interventions: Other: Low Frequency Blood Flow Restriction Training Group
- High Frequency Blood Flow Restriction Training Instability Group (Experimental): Subjects allocated to this group performed squat exercise 6 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM on instability pneumatic discs.
  Interventions: Other: High Frequency Blood Flow Restriction Training Instability Group
- Low Frequency Blood Flow Restriction Training Instability Group (Experimental): Subjects allocated to this group performed squat exercise 3 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM on instability pneumatic discs
  Interventions: Other: Low Frequency Blood Flow Restriction Training Instability Group
- Control Group (Sham Comparator): The subjects of this group performed squat exercise 6 days a week but without BFR. Pneumatic cuff will be wrapped around the thigh of the subjects but it would not be inflated.
  The subjects of this group performed squat exercise 6 days a week but without BFR. Pneumatic cuff were applied to the most proximal part of the thighs and arms but were not inflated.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: High Frequency Blood Flow Restriction Training Group — Subjects allocated to this group performed squat exercise 6 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM.
  Blood flow restriction cuffs were applied to the most proximal part of the thighs and arms. Each subject performed 75 repetitions in total across 4 sets of squats in the order of 30-15-15-15. Rest between sets was 30 sec. Subjects were instructed to tummy tuck while performing the exercise.
  Arms: High Frequency Blood Flow Restriction Training Group
Other: Low Frequency Blood Flow Restriction Training Group — Subjects allocated to this group performed squat exercise 3 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM.
  Blood flow restriction cuffs were applied to the most proximal part of the thighs and arms. Each subject performed 75 repetitions in total across 4 sets of squats in the order of 30-15-15-15. Rest between sets was 30 sec. Subjects were instructed to tummy tuck while performing the exercise.
  Arms: Low Frequency Blood Flow Restriction Training Group
Other: High Frequency Blood Flow Restriction Training Instability Group — Subjects allocated to this group performed squat exercise 6 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM on instability pneumatic discs.
  Blood flow restriction cuffs were applied to the most proximal part of the thighs and arms. Each subject performed 75 repetitions in total across 4 sets of squats in the order of 30-15-15-15. Rest between sets was 30 sec. Subjects were instructed to tummy tuck while performing the exercise.
  Arms: High Frequency Blood Flow Restriction Training Instability Group
Other: Low Frequency Blood Flow Restriction Training Instability Group — Subjects allocated to this group performed squat exercise 3 days per week for 2 weeks with B Strong blood flow restriction cuffs, with the pressure set at 300mmHg of mercury for arm and 350mmHg of mercury for thigh and 30% of 1RM on instability pneumatic discs.
  Blood flow restriction cuffs were applied to the most proximal part of the thighs and arms. Each subject performed 75 repetitions in total across 4 sets of squats in the order of 30-15-15-15. Rest between sets was 30 sec. Subjects were instructed to tummy tuck while performing the exercise.
  Arms: Low Frequency Blood Flow Restriction Training Instability Group
Other: Control Group — The subjects of this group performed squat exercise 6 days a week but without BFR. Pneumatic cuff were applied to the most proximal part of the thighs and arms but were not inflated.
  Each subject performed 75 repetitions in total across 4 sets of squats in the order of 30-15-15-15. Rest between sets was 30 sec. Subjects were instructed to tummy tuck while performing the exercise.
  Arms: Control Group

SUMMARY:
Effects of short duration blood flow restriction training on musculoskeletal and performance outcomes.

DETAILED DESCRIPTION:
Often after 40 years of age due to decrease in physical activity, muscle strength and performance starts gradually declining. However, regular resistance training can decelerate age related decline in musculoskeletal system and it is considered a major contributing factor in optimizing health and longevity. The beneficial effects of resistance training include decreased resting blood pressure, improved lipid profiles, improved glucose metabolism, improved bone mineral density, decreased lower back pain, enhanced flexibility, increased resting metabolic rate, improved maximal aerobic capacity and alleviated symptoms of arthritis.

According to American College of Sports Medicine, at least loads >70% of an individual's one-repetition maximum (1RM) are required to maintain muscle mass and strength. Exercises done with heavy loads of more than >70% of individual 1RM are sometimes referred to traditional resistance training or high-load resistance training (HLRT). However, it is worth mentioning that HLRT may not be suitable for specific populations due to the excessive mechanical stress during exercises on joints and ligaments which may lead to injury. These populations may include novices, individuals recovering from an injury or suffering from chronic diseases, those with disabled limbs as well as the elderly who cannot endure the continual high mechanical stress caused by heavy resistance training.

Alternative training methods to HLRT exists that do not put excessive mechanical loads on the musculoskeletal system, yet can lead to increased muscle mass and strength. One such training method is called blood flow restriction training (BFRT).

In recent years, low load resistance training (< 40% 1RM) combined with blood flow restriction (BFR) has gained much attention as a feasible alternative to HLRT for maintaining or improving muscle mass and strength.

BFR is usually accomplished by inflating a pneumatic cuff or specially designed elastic bands around the most proximal region of the upper and/or lower limbs. Training loads are usually between 20%-40% 1-RM, 75 repetitions per exercise (15- 30 repetitions per set) or sets to failure. During BFRT pressure is applied in such a way that only venous return is blocked while maintaining arterial inflow to the muscles. It causes hypoxia within the muscles. When exercise is performed with BFR, there is an increase in intramuscular pressure beneath the cuff, which further disturbs the blood flow.

Although the use of BFRT seems very enticing and a viable alternative to HLRT but the mechanisms underpinning the hypertrophic adaptations are yet to be fully determined. Over the years numerous theories have been put forth but general consensus of scientific community is that during BFRT, metabolic stress from vascular occlusion and mechanical tension from resistance training may lead to synergistic increases in muscle hypertrophy and strength. At a cellular level, metabolites accumulation like lactate and reactive oxygen species, hormonal differences, cell-to-cell signaling, cellular swelling, and intracellular signaling pathways have all been proposed.

Metabolites, which accumulate during exercise that are known mediators of muscular hypertrophy, are amplified by BFR's relative ischemic and hypoxic conditions. They are believed to induce earlier, peripherally mediated fatigue, resulting in greater motor unit recruitment, as suggested by the fact that BFRT has similar recruitment to that of HLRT. In addition, type II fast-twitch muscle fibers are activated during BFRT.

The benefits of BFRT may also be partially explained by the proliferation and activation of satellite cells (multipotent cells within muscle connective tissue responsible for muscle growth and regeneration) due to increased production of reactive oxygen species such as nitric oxide results from fluctuations in oxygen availability.

BFRT can be performed in either low frequency or high frequency. For low frequency, it is recommended to perform BFRT 2-3 times per week and the intervention lasts longer than three weeks. For high frequency, it is recommended to perform BFRT less than 3 weeks 1-2 times per day. High-frequency BFRT can be potentially useful for clinicians since the technique can provide positive physiological adaptations in short terms.

There are numerous studies conducted on short duration high frequency (<3 weeks intervention) BFRT. The duration of the intervention ranges between 1-3 weeks and frequency of training sessions ranges from 6-16 sessions per week to 24 sessions in 3 weeks. Short duration BFRT studies have positive effects on muscle strength, muscle size, performance, hormonal levels, inflammatory marks and satellite cells. However, there are still research gaps that needs to be addressed.

Difference between the effects of varied frequency short duration BFRT protocols i.e., high frequency vs low frequency on musculoskeletal and performance outcomes is still unclear. Furthermore, limited studies have been conducted on the effect of BFRT on muscles proximal to the BFR site. Often the studies have focused on chest and shoulder muscles but have reported conflicting results. One study assessed the effects of lower limb BFRT on trunk muscles (gluteus maximus, iliopsoas and lumber L4-5) however, it reported that BFR walk training does increase muscle mass in the trunk muscles.

To the best of our knowledge no study has assessed the effects of lower limb BFRT on abdominal muscles. Furthermore, research has shown that instability training can enhance abdominal muscles activation. However, effects of addition of instability during BFRT on musculoskeletal and performance outcomes are not known. Therefore, this study is designed to address some of the current research gaps that exists in BFRT protocols. This study will compare the effects of short duration BFRT protocols (high frequency vs low frequency) on musculoskeletal and performance outcomes. Furthermore, this study will try to understand the effects of addition of instability during BFRT on abdominal muscles.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary males (< 2.5h/week physical activity) or < 300 METs per week (36)
* Age 18-30 years
* BMI between 18.5-29.9
* Free from any lower-limb pain or injury
* No previous experience with BFRT
* Ankle brachial index values between 0.9-1.4
* Not doing regular strength training of lower limb in the past 6 months
* No strenuous physical activities 72h before and during the study period
* Non-smokers

Exclusion Criteria:

* Any injuries of the musculoskeletal system that could prevent the participants from training or testing
* Any use of medication and/or supplements (e.g., protein powder, vitamins, creatine, NSAIDs, etc.)
* Peripheral arterial disease
* Diabetes and hypertensive patients

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-07-08 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Thigh Muscles Ultrasound Assessment | 2 weeks
  Subject lying in supine position. 50% of thigh length was measured from ASIS to mid patella. Ultrasound measurements of muscle thickness of bilateral rectus femoris, and vastus intermedius were performed.
Abdomen Muscles Ultrasound Assessment | 2 weeks
  Subject lying in supine position. The images of bilateral, transverse abdominis, internal oblique and external oblique were taken by placing the probe transversely in the mid-axillary line, between the subcostal line and the iliac crest 15 cm lateral to the umbilicus. For the rectus abdominis examination, the probe was placed transversely 3 cm lateral to the umbilicus.
Thigh Muscles Strength Assessment | 2 weeks
  Subject sitting on a table unsupported. Knee in 75° flexion. Dynamometer was fixed with the table with the help of a strap the other end of the strap was fixed with subject's leg just above the ankle joint. Patient performed MVC for 5 seconds. First 2 seconds submaximal effort. Last 3 seconds maximum effort. 3 trials. 2 mins break between the trails.
Abdominal Muscles Strength Assessment | 2 weeks
  Subject stood in a custom made frame. Knee slightly bent. Heels on the mark so it is standardized for all subjects. Knees and thighs secured and tightened with belt. Chest harness placed and connected to the dynamometer belt. Subject was positioned in 17.5° trunk flexion. Trunk angle checked with goniometer. Patient performed MVC for 5 seconds. First 2 seconds submaximal effort. Last 3 seconds maximum effort. 3 trials. 2 mins break between the trails.
Thigh Muscles Electromyography Assessment | 2 weeks
  Subject sitting on a table unsupported. Knee in 75° flexion. For quadriceps muscles the electrodes were placed approximately half the distance between the knee and the iliac spine.Patient performed MVC for 5 seconds. First 2 seconds submaximal effort. Last 3 seconds maximum effort. 3 trials. 2 mins break between the trails.
Abdominal Muscles Electromyography Assessment | 2 weeks
  Subject stood in a custom made frame. Knee slightly bent. Heels on the mark so it is standardized for all subjects. Knees and thighs secured and tightened with belt. Chest harness placed and connected to the dynamometer belt. Subject was positioned in 17.5° trunk flexion. For rectus abdominis the electrodes were placed 3 cm lateral to the umbilicus. For external oblique the electrodes were placed 15 cm lateral to the umbilicus. Patient performed MVC for 5 seconds. First 2 seconds submaximal effort. Last 3 seconds maximum effort. 3 trials. 2 mins break between the trails.
Jump Assessment | 2 weeks
  Subjects were standing 2 meters away from the mobile stand. My jump 3 mobile app was used for assessment. For jump assessment the mobile was fixed on a stand and placed in front of the subject.

SECONDARY OUTCOMES:
Delayed Onset Muscle Soreness Assessment | 2 weeks
  Quadriceps palpated with two fingers on five different locations of bilateral legs: distal, middle, and proximal parts of the rectus femoris, vastus lateralis, and vastus medialis muscles. The measurement locations recorded on transparent, acetate paper. Palpations done in a standing position and subjects familiarized to apply palpation pressures two times before the baseline measurements.
Rating of Perceived Exertion Scale | 2 weeks
  Rating of perceived exertion scale was used to identify the patients' intensity of exercise. It is a numerical scale that ranges from 1 to 10, where 1 means "no exertion at all" and 10 means "maximal exertion."

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, Study Chair — asghar.khan@riphah.edu.pk; Waqar Ahmed Awan, PhD, Study Chair — Riphah International University; Saad Rauf, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No